CLINICAL TRIAL: NCT01969994
Title: A Single-Center, Open-Label Study to Evaluate the Absorption, Metabolism, and Excretion of (-)-[2-14C]Epicatechin Following Oral Intake
Brief Title: Absorption, Metabolism, and Excretion of (-)-[2-14C]Epicatechin in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Institutes for Pharmaceutical Discovery, LLC (Industry)
Collaborators: Covance (Industry); Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 8215022
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: ADME
Keywords: Epicatechin; Flavanols; Procyanidins; Polyphenols; Phytonutrients; AMDE; Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Controlled dietary background & (-)-[2-14C]epicatechin intake (Experimental)
  Interventions: Other: Controlled dietary background; Other: (-)-[2-14C]epicatechin intake

INTERVENTIONS:
Other: Controlled dietary background — Controlled dietary flavanol-/procyanidin- background, consisting of daily intake for 14 days (day -17 to -4) of a commercially available flavanol-/procyanidin-containing cocoa-based drink (250 mg cocoa flavanols; 40 mg of (-)-epicatechin) followed by a 4-day period (day -4 to 0) of a low-flavanol diet.
Other: (-)-[2-14C]epicatechin intake — Single oral intake of an aqueous solution of a mixture of non-radiolabeled (-)-epicatechin and a single-carbon-14 radiolabeled (-)-[2-14C]epicatechin. The target amount of EC delivered with test drink will be 60 mg, 58.5 mg of which consist of non-radiolabled EC and 1.54 mg (300 µCi) consist of (-)-[2-14C]epicatechin.
  Other Names: (-)-cis-3,3',4',5,7-Pentahydroxyflavane; (2R,3R) - 2- (3,4- Dihydroxyphenyl) - 3,4- dihydro- 1(2H) - benzopyran- 3,5,7- triol

SUMMARY:
The purpose of this study is to determine the absorption, metabolism and excretion of (-)-epicatechin using the radiolabeled tracer (-)-[2-14C]epicatechin in healthy male volunteers observing a flavanol-/procyanidin-controlled background diet.

DETAILED DESCRIPTION:
Flavanols and their oligomeric derivatives, the procyanidins, are plant-derived compounds commonly present in the human diet. Accumulating data demonstrate a causal role for dietary flavanols in mediating the cardiovascular benefits associated with the consumption of flavanol-/procyanidin-containing foods. In this context, there exists a great interest in understanding the absorption, distribution, metabolism and excretion (ADME) of flavanols in humans. While significant advances in understanding the ADME of flavanols were made, the data obtained thus far remain fairly preliminary and with significant shortfalls and seeming contradictions. Aimed at addressing the challenges and gaps of previous investigations, this study will investigate the ADME of (-)-epicatechin, one of the most abundant dietary flavanols, following the intake of radiolabeled (-)-[2-14C]epicatechin by healthy humans observing a flavanol-/procyanidin-controlled background diet.

ELIGIBILITY:
Inclusion Criteria1.

1. males, in good health, between 18 and 50 years of age and between 60 and 100 kg;
2. body mass index (BMI) between 19 and 30 kg/m2.
3. clinical laboratory evaluations (including clinical chemistry [fasted at least 10 hours], hematology, and urinalysis) within the reference range for the testing laboratory, unless deemed not clinically significant by the Investigator;
4. negative hepatitis panel (including hepatitis B surface antigen [HbsAg] and hepatitis C virus antibody [anti-HCV]) and human immunodeficiency virus (HIV) antibody screens;
5. a minimum of 1 bowel movement per day.

Exclusion Criteria:

1. history or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urological, or psychiatric disorders;
2. allergies to peanuts, nuts, or other foods;
3. lactose intolerance;
4. history of stomach or intestinal surgery, except that appendectomy or hernia were allowed;
5. history of alcoholism or drug addiction within 1 year prior to study entry (ie, at Screening);
6. use of any tobacco products (including cigarette, pipe, cigar, chewing, nicotine patch, or nicotine gum) within 6 months prior to study entry;
7. use of any agents (excluding those provided as part of this study procedure) affecting the liver enzymes;
8. use of aspirin-containing drugs and any other over-the-counter, non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) during the study, unless deemed acceptable by the Investigator;
9. use of any alcohol-containing or caffeine-containing products/medications within 72 hours prior to (-)-[2-14C]epicatechin ingestion;
10. regular consumption of more than 2 alcoholic drinks per day;
11. vegans, vegetarians and/or anyone who consumed less than 1 to 2 servings of fruits and or vegetables per day;
12. participation in more than one other radiolabeled investigational study drug trial within 12 months prior to study entry or exposure to significant radiation within 12 months prior to study entry;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in levels of (-)-[2-14C]epicatechin-derived radioactivity in blood, plasma, urine, and feces; | 0 (prior to the ingestion of (-)-[2-14C]epicatechin), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours postdose, and at every subsequent 24 hour timepoint up to 240 h or until volunteers meet discharge criteria

SECONDARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters of total (-)-[2-14C]epicatechin-derived radioactivity levels in plasma, urine and feces. | 0 (prior to the ingestion of (-)-[2-14C]epicatechin) up to 240 h or untill volunteers meet discharge criteria
  PK parameters: Cmax: maximum observed concentration in plasma; tmax: time to maximum concentration in plasma; AUC0-t: area under the plasma radioactivity-time curve from hour 0 to the last measurable concentration in plasma; AUC0-∞: area under the plasma concentration-time curve extrapolated to infinity; λZ: apparent terminal elimination rate constant in plasma; t1/2: apparent terminal elimination half-life in plasma; CL/F: systemic clearance; Vd/F: apparent volume of distribution; CLR: renal clearance; Aeu(0-t): cumulative amount excreted in the urine over each sampling interval and the total interval examined; Aef(0-t): Cumulative amount excreted in the feces over each sampling interval and the total interval examined.
Composite of pharmacokinetic (PK) parameters of individual (-)-[2-14C]epicatechin metabolites in plasma and urine | 0 (prior to the ingestion of (-)-[2-14C]epicatechin) up to 240 h or untill volunteers meet discharge criteria
  PK parameters of each (-)-epicatechin metabolite:
  Cmax: maximum observed concentration in plasma; tmax: time to maximum concentration in plasma; AUC0-t: area under the plasma concentration-time curve from hour 0 to the last measurable concentration in plasma; AUC0-∞: area under the plasma concentration-time curve extrapolated to infinity; λZ: apparent terminal elimination rate constant in plasma; t1/2: apparent terminal elimination half-life in plasma; CL/F: systemic clearance; Vd/F apparent volume of distribution; CLR: renal clearance; Aeu(0-t): cumulative amount excreted in the urine over each sampling interval and the total interval examined.

CONTACTS AND LOCATIONS:
Overall Officials: Christine L Hale, MD, Principal Investigator — Covance Clinical Pharmacology Inc.; Michael Fare, Study Director — IPD, LLC; Javier I Ottaviani, Ph.D., Study Director — Mars, Inc.
Locations (1):
- Covance Clinical Pharmacology Inc., Madison, Wisconsin, United States

REFERENCES:
- [Derived] Ottaviani JI, Borges G, Momma TY, Spencer JP, Keen CL, Crozier A, Schroeter H. The metabolome of [2-(14)C](-)-epicatechin in humans: implications for the assessment of efficacy, safety, and mechanisms of action of polyphenolic bioactives. Sci Rep. 2016 Jul 1;6:29034. doi: 10.1038/srep29034. PMID 27363516